CLINICAL TRIAL: NCT02570087
Title: Benefits of Chronic Total Coronary Occlusion Percutaneous Intervention in Patients With Chronic Heart Failure and Reduced Ejection Fraction.
Brief Title: Benefits of CTO-PCI in Selected Cases With HFrEF (CTOHFrEF)
Acronym: CTOHFrEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Montserrat Cardona, Consultant, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CTOHFrEF
Record Dates: First submitted 2015-09-25; First posted 2015-10-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Total Occlusion Vessel
Keywords: Coronary ChronicTotal Occlusion; Coronary Angioplasty; Reduced Ejection Fraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Successful CTO PCI (Active Comparator): Successful chronic total coronary occlusion percutaneous intervention (CTO-PCI)
  Interventions: Procedure: chronic total coronary occlusion percutaneous intervention
- Unsuccessful CTO PCI (No Intervention): Unsuccessful chronic total coronary occlusion percutaneous intervention (CTO-PCI)

INTERVENTIONS:
Procedure: chronic total coronary occlusion percutaneous intervention — Percutaneous intervention of chronic total coronary occlusion with stent implantation
  Arms: Successful CTO PCI

SUMMARY:
The investigators studied the effect of CTO-PCI on left ventricular function and clinical parameters in patients with HFrEF.

DETAILED DESCRIPTION:
Observational studies have shown that chronic total coronary occlusion percutaneous intervention (CTO-PCI) improves angina, left ventricular ejection fraction (LVEF), and survival. None of these studies aimed to assess the benefits in populations with heart failure with reduced ejection fraction (HFrEF). The investigators studied the effect of CTO-PCI on left ventricular function and clinical parameters in patients with HFrEF.

Using cardiac magnetic resonance (CMR), the investigators studied 29 patients with HFrEF and evidence of viability and/or ischemia in the territory supplied by an occluded vessel who were successfully treated with CTO-PCI. Non-CTO PCI was also performed in patients with multi-vessel disease, . Imaging parameters, clinical status, and brain natriuretic peptide (BNP) levels were evaluated before and six months after CTO-PCI.

ELIGIBILITY:
Inclusion Criteria:

* At least one chronic total coronary occlusion
* LVEF ≤40% by CMR
* Evidence of myocardial viability and/or ischemia in at least two contiguous segments subtended by the occluded vessel.

Exclusion Criteria:

* Women of childbearing age or pregnant
* Claustrophobia
* Admission to hospital within the previous 90 days due to decompensated heart failure, myocardial infarction or unstable angina.
* Severe valvulopathy
* Pacemaker or implantable cardioverter defibrillator
* Indication for coronary artery bypass surgery
* Heart transplantation waiting list
* Follow-up not feasible
* Life expectancy shorter than 12 months.
* Iodine contrast or gadolinium allergy
* Aspirin or clopidogrel allergy
* Asthma
* NYHA IV class
* Liver cirrosis
* Noncompliance with medical treatment
* Chronic kidney disease with serum creatinine levels ≥ 2.5 mg/dl or glomerular filtration rate ≤30 ml/min/1.73m2
* Evidence of active bleeding
* High risk of bleeding
* CTO distal vessel not visible through collateral circulation
* CTO distal vessel diameter <2mm
* Absence of acceptable vascular access

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-07; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (%) | 6 months
  Evaluate changes in left ventricular function by cardiac magnetic resonance imaging 6 months after CTO PCI

SECONDARY OUTCOMES:
NYHA functional class (I-V) | 6 months
  Evaluate changes in NYHA functional class 6 months after CTO PCI
Myocardial ischemia | 6 months
  Evaluate changes in number of segments with induced ischemia by cardiac magnetic resonance imaging 6 months after CTO PCI
Brain Natriuretic Peptide (pg/ml) | 6 months
  Evaluate changes in brain natriuretic peptide 6 months after CTO PCI
Incidence of in-hospital CTO PCI major adverse events | 6 months
  Safety evaluation of CTO PCI in patients with HFrEF (periprocedural mortality, periprocedural STEMI or need for urgent myocardial revascularization surgery)

REFERENCES:
- [Derived] Cardona M, Martin V, Prat-Gonzalez S, Ortiz JT, Perea RJ, de Caralt TM, Masotti M, Perez-Villa F, Sabate M. Benefits of chronic total coronary occlusion percutaneous intervention in patients with heart failure and reduced ejection fraction: insights from a cardiovascular magnetic resonance study. J Cardiovasc Magn Reson. 2016 Nov 5;18(1):78. doi: 10.1186/s12968-016-0287-5. PMID 27814739